CLINICAL TRIAL: NCT03482219
Title: Rehabilitation for Arm Coordination and Hand Movement in Systemic Sclerosis (The REACH Study)
Brief Title: Rehabilitation for Arm Coordination and Hand Movement in Systemic Sclerosis
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Scleroderma Foundation (Unknown)
Responsible Party: Principal Investigator, Susan Murphy, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00141111
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Systemic Sclerosis; SSc
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive treatment (Experimental): Participants will undergo 8 sessions with an occupational therapist. Participants will meet with the occupational therapist to establish the home exercise program and set up the home exercise app. The app has videos depicting each exercise and ability to track adherence to exercises. The occupational therapy consists of the following which will be provided as appropriate:
  1. Thermal Modalities Hot packs, focused on areas with limitations Paraffin, focused on digital limitations
  2. Application of the Physiotouch (a low-intensity negative pressure device)
  3. Passive Range of Motion
  4. Active Range of Motion
  5. Functional Activities
  Interventions: Other: Occupational therapy; Other: Home app intervention
- Home app intervention (Active Comparator): Participants will meet with the occupational therapist to establish the home exercise program and set up the home exercise app. The app has videos depicting each exercise and ability to track adherence to exercises.
  Interventions: Other: Home app intervention

INTERVENTIONS:
Other: Occupational therapy — The Occupational therapy intervention includes various thermal modalities, manual therapy, Physiotouch (Healthy Life Devices Ltd) and education. The home app intervention involves one session of education with the occupational therapist.
  Arms: Intensive treatment
Other: Home app intervention — The app consists of videos depicting each exercise and ability to track adherence to exercises.

SUMMARY:
The purpose of this study is to test two rehabilitation programs to improve arm function for patients with scleroderma. This is a Phase 2 randomized controlled trial in which participants will be assessed at baseline, 8 weeks, and 18 weeks. Participants will be randomized into an intensive intervention (8 individual sessions of occupational therapy plus a home exercise app) versus a home app treatment alone. The results of this study will be used to design a large multi-site trial in which optimized rehabilitation strategies can be used to help patients improve their arm function.

DETAILED DESCRIPTION:
The specific aims of this study are to:

1. Determine the short and longer-term effects of an intensive (8-week in-person occupational therapy treatment with prescribed home exercises) on improving arm function versus home exercise alone.

   This study's hypothesis is that immediately following treatment at 8 weeks and at 18 weeks, participants randomized to the in-person occupational therapy will have significant improvements in the QuickDASH disability measure, PROMIS physical function measure, and total active hand function compared to the home exercise alone.
2. Determine how adherence to home exercise in both groups influences treatment effects.

This study's hypothesis is that adherence will independently predict improvement in outcomes at 8 and 18 weeks regardless of treatment group assignment and that higher adherence to the home exercise program will result in greater and more long-lasting improvements.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of systemic sclerosis including:

  * Diffuse cutaneous subset
  * Disease duration < 5 years from 1st non Raynaud phenomenon sign or symptom
* Have a contracture of the hand and other joint in at least one arm, such as wrist, elbow, or shoulder, with the ability to demonstrate active range of motion in that arm
* Willing to travel to participate in therapy and outcome assessments.
* Have an Android, iPhone, iPad or computer tablet to load the home exercise App.
* English speaking

Exclusion Criteria:

* issues that preclude meaningful participation in study procedures (e.g. concurrent or complex medical issues, inability to use home exercise app, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
quickDASH | Change from Baseline at 8 weeks and 18 weeks
  self-report questionnaire of physical function and symptoms. This is an 11-item questionnaire in which difficulty in several tasks involving the upper extremity are rated as well as interference and severity of symptoms. Items are averaged and converted to a 0 - 100 scale; a higher score indicates worse function.

SECONDARY OUTCOMES:
Physical Function | Change from Baseline at 8 weeks and 18 weeks
  PROMIS physical function 8-item short form. The US population mean score for this measure is 50 with SD of 10, and a higher score denotes better function
Total Hand Function | Change from Baseline at 8 weeks and 18 weeks
  Summary score of degrees of active range of motion in hand. This is calculated by summing the total active range of motion for each finger and thumb by goniometer (260 degrees in each finger and 135 in the thumb). A total score of 1125 is possible and a higher score equals more range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Susan Murphy, ScD OTR, Principal Investigator — Associate Professor
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy SL, Barber M, Huang S, Sabbagh M, Cutter G, Khanna D. Intensive and app-delivered occupational therapy to improve upper extremity function in early diffuse cutaneous systemic sclerosis: a pilot two-arm trial. Rheumatology (Oxford). 2021 Nov 3;60(11):5002-5011. doi: 10.1093/rheumatology/keab339. PMID 33839775